CLINICAL TRIAL: NCT03436290
Title: Surgery for Cancer With Option of Palliative Care Expert: A Randomized Trial of an Early Palliative Care Intervention for Patients Undergoing Surgery for Cancer
Brief Title: Surgery for Cancer With Option of Palliative Care Expert
Acronym: SCOPE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Myrick C. Shinall, Jr., MD, PhD, Assistant Professor of Surgery, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SCOPE
Record Dates: First submitted 2017-12-28; First posted 2018-02-19 (Actual); Results first posted 2024-06-10 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2025-12

CONDITIONS: Cancer
Keywords: Palliative Care
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Palliative Care Intervention (Experimental)
  Interventions: Behavioral: Palliative Care Intervention
- Standard of Care (No Intervention)

INTERVENTIONS:
Behavioral: Palliative Care Intervention — These patients will receive the palliative care intervention.
  Arms: Palliative Care Intervention

SUMMARY:
Frequently people diagnosed with cancer experience physical and emotional symptoms during the course of their disease. These symptoms can be very distressing to both the patient and the family members. The study doctor wants to know if the introduction of a team of clinicians that specialize in the lessening of many of these distressing symptoms may improve your overall care. This team of clinicians is called the palliative care team and they focus on ways to improve your pain and other symptom management (i.e. shortness of breath, fatigue, anxiety, etc.) and to assist you and your family in coping with the emotional, social, and spiritual issues associated with your diagnosis. The team consists of physicians, advanced practice nurses, case managers, and nurses who have been specially trained in the care of patients facing serious illness.

This research study is being done because although many people with cancer receive palliative care late in the course of their illness, the study team thinks palliative care may be more useful when it is started earlier and in this case before surgery. The main purpose of this study is to compare two types of care -usual surgery and cancer care and usual surgery and cancer care with comprehensive palliative care services to see which is better for improving the experience of patients and families with cancer.

DETAILED DESCRIPTION:
The Surgery for Cancer with Option of Palliative Care Expert (SCOPE) Trial is an investigation that will study the effect of a palliative care implementation during the preoperative, perioperative, and postoperative phase for adults undergoing cancer surgery for selected gastrointestinal and genitourinary malignancies. SCOPE will be a single-blind, single-institution randomized controlled trial of 236 patients. Intervention arm patients will receive a preoperative outpatient specialty palliative care consultation from a palliative care provider (physician or nurse practitioner) in addition to inpatient and outpatient palliative care follow-up postoperatively. Control arm patients will receive usual care with palliative care available at the discretion of the primary treatment team (currently these patients rarely get palliative care and usually only in the last weeks of life). The central hypothesis of the SCOPE Trial is that preoperative, perioperative, and postoperative specialty palliative care will improve patient functioning and quality of life in patients undergoing resection of selected GI and GU malignancies.

ELIGIBILITY:
Inclusion Criteria:

adult patients (≥18 years old) scheduled for one of the following abdominal operations with intent to provide cure or durable oncologic control of malignancy:

1. Total or partial gastrectomy requiring anastomosis
2. Total or partial pancreatectomy
3. Partial hepatectomy
4. Colectomy or proctactomy if one of the following 3 conditions is also met:

   i) patient age is 65 years or older ii) disease is metastatic iii) disease is locally invasive requiring extensive resection
5. Radical cystectomy
6. Pelvic exenteration
7. Abdominal debulking for ovarian or endometrial carcinoma
8. Cytoreductive surgery and hyperthermic intraperitoneal chemotherapy

Exclusion Criteria:

1. Non-English speaking patient
2. Residence >150 miles away from Vanderbilt and do not visit the Nashville area regularly
3. No telephone or otherwise unwilling/unable to complete follow-ups
4. Prisoner
5. Current enrollment in a study that does not allow co-enrollment or that uses a non-pharmacologic, non-procedural intervention directed at surgical or cancer care.
6. Deaf
7. Severe prior cognitive or neurodegenerative disorder that prevents a patient from living independently at baseline
8. Inability to obtain informed consent from patient meeting all inclusion criteria for the following reasons:

   1. Attending surgeon refusal
   2. Patient refusal
   3. Period of time between screening patient and time of operation does not allow preoperative outpatient palliative care visit.
9. Currently participating in palliative care or seeing a palliative care provider.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 236 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2022-02-24 (Actual); Study Completion 2026-11 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Myrick C Shinall, MD, Principal Investigator — Assistant Professor
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Shinall MC Jr, Martin SF, Karlekar M, Hoskins A, Morgan E, Kiehl A, Bryant P, Orun OM, Raman R, Tillman BF, Hawkins AT, Brown AJ, Bailey CE, Idrees K, Chang SS, Smith JA Jr, Tan MCB, Magge D, Penson D, Ely EW. Effects of Specialist Palliative Care for Patients Undergoing Major Abdominal Surgery for Cancer: A Randomized Clinical Trial. JAMA Surg. 2023 Jul 1;158(7):747-755. doi: 10.1001/jamasurg.2023.1396. PMID 37163249
- [Derived] Orun OM, Shinall MC Jr, Hoskins A, Morgan E, Karlekar M, Martin SF, Ely EW, Raman R. Statistical analysis plan for the Surgery for Cancer with Option of Palliative Care Expert (SCOPE) trial: a randomized controlled trial of a specialist palliative care intervention for patients undergoing surgery for cancer. Trials. 2021 Apr 29;22(1):314. doi: 10.1186/s13063-021-05256-y. PMID 33926535
- [Derived] Shinall MC Jr, Hoskins A, Hawkins AT, Bailey C, Brown A, Agarwal R, Duggan MC, Beskow LM, Periyakoil VS, Penson DF, Jarrett RT, Chandrasekhar R, Ely EW. A randomized trial of a specialist palliative care intervention for patients undergoing surgery for cancer: rationale and design of the Surgery for Cancer with Option of Palliative Care Expert (SCOPE) Trial. Trials. 2019 Dec 11;20(1):713. doi: 10.1186/s13063-019-3754-0. PMID 31829237

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard of Care: Patients received standard perioperative care
Period: Overall Study
Arm/Group | Palliative Care Intervention | Standard of Care
Started | 118 | 118
Completed | 77 (Number who received all elements of the intervention per protocol) | 118
Not Completed | 41 | 0
Not completed — Post-randomization Exclusion | 1 | 0
Not completed — Death | 6 | 0
Not completed — Withdrawal by Subject | 4 | 0
Not completed — Protocol Violation | 30 | 0

BASELINE CHARACTERISTICS:
Population: Excludes one patient who was excluded after randomization
Groups:
- Standard of Care: These patients received standard perioperative care
- Total: Total of all reporting groups
Arm/Group | Palliative Care Intervention | Standard of Care | Total
Number analyzed (Participants) | 117 | 118 | 235
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 62.3 [56.6 to 69.3] | 66.6 [57.8 to 71.6] | 65 [56.8 to 71.1]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 48 | 94
  Male | 71 | 70 | 141
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 117 | 116 | 233
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 4 | 9
  White | 111 | 113 | 224
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 117 | 118 | 235
FACT-TOI [Median (Inter-Quartile Range); unit: units on a scale] — FACT-Gastric Trial Outcome Index (TOI) is an efficient summary index of physical/functional outcomes and is comprised of two subscales from the FACT-Gastric Score: the physical wellbeing subscale (7 questions) and the functional wellbeing scale (7 questions). Each question uses a 5-point Likert scale ranging from 0 (Not at all) to 4 (Very much). Total scores on the FACT-TOI range from 0-56. The higher the score, the better the quality of life.
  units on a scale | 43.0 [34.8 to 50.0] | 44.0 [38.0 to 51.0] | 43.0 [36.0 to 50.0]
FACT-G [Median (Inter-Quartile Range); unit: units on a scale] — The FACT-G is a patient self-administered 27-item questionnaire that measures health state in cancer patients in prior 7 days, including physical, social, emotional, and functional well-being. Scoring: Five-point scale: 0 (not at all) to 4 (very much). Total score is from 0-108. The higher the score, the better quality of life (QOL).
  units on a scale | 85.0 [72.9 to 94.0] | 87.4 [76.0 to 95.0] | 86.0 [74.8 to 94.6]

OUTCOME MEASURES:

1. Primary Outcome: Physical and Functional Quality of Life as Measured by the FACT-G TOI
Description: FACT-Gastric Trial Outcome Index (TOI) is an efficient summary index of physical/functional outcomes and is comprised of two subscales from the FACT-Gastric Score: the physical wellbeing subscale (7 questions) and the functional wellbeing scale (7 questions). Each question uses a 5-point Likert scale ranging from 0 (Not at all) to 4 (Very much). Total scores on the FACT-TOI range from 0-56. The higher the score, the better the quality of life.
Time Frame: 90 days after operation
Population: Includes all patients who completed the FACT-G instrument at 90 days
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Palliative Care Intervention | Standard of Care
Number analyzed (Participants) | 104 | 113
units on a scale | 45.0 [36.2 to 50.0] | 45.0 [39.0 to 50.0]

2. Secondary Outcome: Quality of Life as Measured by the FACT-G
Description: The FACT-G is a patient self-administered 27-item questionnaire that measures health state in cancer patients in prior 7 days, including physical, social, emotional, and functional well-being. Scoring: Five-point scale: 0 (not at all) to 4 (very much). Total score is from 0-108. The higher the score, the better quality of life (QOL).
Time Frame: 90 days after operation
Population: All patients who completed the FACT-G instrument at 90 days
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Palliative Care Intervention | Standard of Care
Number analyzed (Participants) | 104 | 113
units on a scale | 88.0 [72.8 to 99.0] | 91.0 [79.5 to 98.3]

3. Secondary Outcome: Days Alive at Home Without an Emergency Room Visit
Description: A count of all the days that the patient 1) has no emergency room visits, and 2) is not an inpatient of a hospital or other health-care facility
Time Frame: 90 days after operation
Population: All included patients
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Palliative Care Intervention | Standard of Care
Number analyzed (Participants) | 117 | 118
days | 84 [76 to 86] | 83 [79 to 85]

4. Secondary Outcome: Post-Traumatic Stress Disorder (PTSD) Symptoms
Description: Score on the PTSD Checklist-Civilian Version--a 17-item scale scored from 17-85 with higher scores indicating more PTSD symptoms
Time Frame: 180 days after operation
Reporting Status: Not Posted

5. Secondary Outcome: Overall Survival
Time Frame: 1 year
Population: All included patients
Measure: Number (95% Confidence Interval); unit: proportion of patients surviving 1 year
Arm/Group | Palliative Care Intervention | Standard of Care
Number analyzed (Participants) | 117 | 118
proportion of patients surviving 1 year | 0.83 [0.76 to 0.90] | 0.82 [0.75 to 0.90]

6. Other Pre Specified Outcome: Physical and Functional Quality of Life
Description: FACT-G TOI Score
Time Frame: 180 days, 12 months, 18 months, 24 months, 30 months, 36 months after operation
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Functional Status
Description: Karnofsky Performance Status--a score that ranges from 0 to 100, with 100 indicating full functional status and 0 indicating death
Time Frame: 90 days, 180 days, 12 months, 18 months, 24 months, 30 months, 36 months after operation
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Quality of Life
Description: FACT-G Score
Time Frame: 180 days, 12 months, 18 months, 24 months, 30 months, 36 months after operation
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Depression
Description: PROMIS Depression-6 Score--A six item scale with scores from 5-30 with higher scores indicating more symptoms of depression
Time Frame: 90 days, 180 days after operation
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Anxiety
Description: PROMIS Anxiety-6 Score--A six item scale with scores from 5-30 with higher scores indicating more anxiety
Time Frame: 90 days, 180 days after operation
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Time to Adjuvant Therapy
Description: Number of days from operation until adjuvant chemotherapy or radiation is initiated
Time Frame: 90 days
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Satisfaction With Hospital Stay
Description: The answer to the following question: Using any number from 0 to 10, where 0 is the worst hospital possible and 10 is the best hospital possible, what number would you use to rate this hospital during your stay?
Time Frame: 30 days
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Post-Traumatic Growth
Description: Post-Traumatic Growth Inventory score--a 21-item scale scored from 0-105 with higher scores indicating more growth after trauma
Time Frame: 180 days
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Care-Giver Burden
Description: Zarit Burden Interview score--a 12 item scale with score 0-48 with higher scores indicating more care-giver burden
Time Frame: 90 days, 180 days, 12 months, 18 months, 24 months, 30 months, 36 months after operation
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Hospital Admissions
Description: Number of hospital admissions
Time Frame: 3 years
Reporting Status: Not Posted

16. Other Pre Specified Outcome: ER Visits
Description: Number of visits to the emergency room
Time Frame: 3 years
Reporting Status: Not Posted

17. Other Pre Specified Outcome: Employment
Description: Patient report of whether or not he or she is currently employed (yes/no question) and if yes, whether the employment is full-time or part-time
Time Frame: 180 days, 12 months, 18 months, 24 months, 30 months, 36 months after operation
Reporting Status: Not Posted

18. Other Pre Specified Outcome: Community vs. Facility Residence
Description: Patient report of whether he or she lives in a private residence or in a healthcare facility (i.e. assisted living, long-term care facility, nursing home, etc.)
Time Frame: 180 days, 12 months, 18 months, 24 months, 30 months, 36 months after operation
Reporting Status: Not Posted

19. Other Pre Specified Outcome: Size of Life Space
Description: Life Space Assessment Questionnaire score--a five item scale with scores from 0-120 with higher scores indicating larger life space i.e. larger area traversed during daily activities
Time Frame: 180 days, 12 months, 18 months, 24 months, 30 months, 36 months after operation
Reporting Status: Not Posted

20. Other Pre Specified Outcome: Length of Hospice Enrollment
Time Frame: last 30 days of life
Reporting Status: Not Posted

21. Other Pre Specified Outcome: Receipt of Chemotherapy in Last 14 Days of Life
Time Frame: last 14 days of life
Reporting Status: Not Posted

22. Other Pre Specified Outcome: Days at Home Without an ER Visit in Last 30 Days of Life
Time Frame: last 30 days of life
Reporting Status: Not Posted

23. Other Pre Specified Outcome: Quality of End-of-life Care
Description: FATE-S score
Time Frame: last 30 days of life
Reporting Status: Not Posted

24. Other Pre Specified Outcome: Location of Death
Description: Care-giver report of whether patient died in a private residence or in a healthcare facility such as a nursing home, hospital, or inpatient hospice facility
Time Frame: last 30 days of life
Reporting Status: Not Posted

25. Other Pre Specified Outcome: Survival
Time Frame: 3 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 12 months
Description: As described in the clinical trials.gov definitions
Arm/Group | Palliative Care Intervention | Standard of Care
All-Cause Mortality (participants affected / at risk) | 6/117 | 4/118
Serious Adverse Events (participants affected / at risk) | 0/117 | 0/118
Other Adverse Events (participants affected / at risk) | 0/117 | 0/118

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-02): https://cdn.clinicaltrials.gov/large-docs/90/NCT03436290/Prot_SAP_000.pdf